CLINICAL TRIAL: NCT02440009
Title: A Randomized Trial of Itraconazole in Acute Stages of Allergic Bronchopulmonary Aspergillosis
Acronym: RIA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Professor, Department of Pulmonary Medicine, Principal Investigator, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Histo-15-IMEC-313
Record Dates: First submitted 2015-05-01; First posted 2015-05-12 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Allergic Bronchopulmonary Aspergillosis
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary | interventions — Itraconazole; Azoles; Glucocorticoids; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucocorticoid group (Active Comparator): Oral prednisolone 0.5 mg/kg/day for 4 weeks; 0.25 mg/kg/day for 4 weeks; 0.125 mg/kg/day for 4 weeks. Then taper by 5 mg every 4 weeks and discontinue by the end of 4 months. Patients will also receive inhaled formoterol/fluticasone (6/125 mcg) 1 puff BD and as needed as per the SMART approach for control of asthma
  Interventions: Drug: Glucocorticoids
- Itraconazole plus glucocorticoid group (Experimental): Oral itraconazole 200 mg BD for 6 months AND oral prednisolone 0.5 mg/kg/day for 4 weeks; 0.25 mg/kg/day for 4 weeks; 0.125 mg/kg/day for 4 weeks. Then taper by 5 mg every 4 weeks and discontinue by the end of 4 months. Patients will also receive inhaled formoterol/fluticasone (6/125 mcg) 1 puff BD and as needed as per the SMART approach for control of asthma.
  Interventions: Drug: Itraconazole; Drug: Glucocorticoids

INTERVENTIONS:
Drug: Itraconazole — Oral itraconazole 200 mg BD for 6 months
  Other Names: Azole
  Arms: Itraconazole plus glucocorticoid group
Drug: Glucocorticoids — Oral prednisolone 0.5 mg/kg/day for 4 weeks; 0.25 mg/kg/day for 4 weeks; 0.125 mg/kg/day for 4 weeks. Then taper by 5 mg every 4 weeks and discontinue by the end of 4 months.
  Other Names: Steroid

SUMMARY:
The study evaluates the addition of itraconazole to glucocorticoids in management of acute stages of allergic bronchopulmonary aspergillosis (ABPA). Half of the participants will receive glucocorticoids while the other half will receive itraconazole and glucocorticoids

DETAILED DESCRIPTION:
The management of allergic bronchopulmonary aspergillosis (ABPA) includes two important aspects namely institution of immunosuppressive therapy in the form of glucocorticoids to control the immunologic activity, and close monitoring for detection of relapses. Another possible target is to use antifungal agents to attenuate the fungal burden secondary to the fungal colonization in the airways. Oral corticosteroids are currently the treatment of choice for ABPA associated with bronchial asthma. They not only suppress the immune hyperfunction but are also anti-inflammatory.

Itraconazole, an oral triazole with relatively low toxicity, is active against Aspergillus spp. in vitro and in vivo. The activity of itraconazole against Aspergillus spp. is more than that of ketoconazole. The administration of itraconazole can eliminate Aspergillus in the airways and can theoretically reduce the allergic responses in ABPA. We hypothesize that itraconazole when given in the acute stages of ABPA will decrease the chances of relapse and progression to glucocorticoid-dependent ABPA.

ELIGIBILITY:
Inclusion Criteria:

Treatment naive patients of allergic bronchopulmonary aspergillosis (ABPA) defined by the presence of all the following:

* asthma
* immediate cutaneous hyperreactivity on Aspergillus skin test or A.fumigatus specific IgE levels >0.35 kUA/L
* elevated total IgE levels >1000 IU/mL and, two of the following features:
* presence of precipitating antibodies against A.fumigatus in serum
* fixed or transient radiographic pulmonary opacities
* total eosinophil count >1000/µL
* bronchiectasis on HRCT chest

Exclusion Criteria:

* Intake of systemic glucocorticoids for more than three weeks in the preceding six months
* Exposure to azoles in the last six months
* Immunosuppressive states such as uncontrolled diabetes mellitus, chronic renal failure, chronic liver failure and others
* Patient on immunosuppressive drugs
* Pregnancy
* Enrollment in another trial of ABPA
* Failure to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Relapse rates | 12 months
  Doubling of the baseline IgE levels irrespective of the patient's symptoms or appearance of radiologic infiltrates; or clinical and/or radiological worsening with 50% increase in IgE over the previous baseline value
Glucocorticoid-dependent ABPA | 24 months
  If the patient has relapse on two or more consecutive occasions within 6 months of stopping treatment or requires oral steroids for control of asthma

SECONDARY OUTCOMES:
Proportion of patients with a response rates | Six weeks
Percentage decline in IgE | Six weeks
Time to first relapse | Two years
Treatment-related adverse effects | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Chest Clinic, PGIMER, Chandigarh, India